CLINICAL TRIAL: NCT05887440
Title: Effects of Isokinetic Strength Training of Knee Flexor and Extensor Muscles on Walking in Hemiparetic Patients With Knee Extension Thrust
Brief Title: Isokinetic Strength Training in Hemiparetic Patient With Knee Extension Thrust
Acronym: ISOWALK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 35RC20_9899_ISOWALK
Record Dates: First submitted 2023-04-14; First posted 2023-06-02 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Hemiparesis/Hemiplegia (One Sided Weakness/Paralysis); Gait Disorder
Keywords: Stroke; Extensor thrust; resistance training; Isokinetic; walking speed; rehabilitation
MeSH Terms: conditions — Paresis; Hemiplegia; Mobility Limitation; Stroke

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design (SCED)
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention neither subjects nor staff can be blinded to allocation. The outcome assessors and data analyst will be blinded to research aims and randomization (multiple baseline design before introducing isokinetic strength training)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3 assessments (Experimental): The randomisation provides for 3 assessments of baseline
  Interventions: Behavioral: isokinetic strength training of knee extensor and flexor muscles
- 4 assessments (Experimental): The randomisation provides for 4 assessments of baseline
  Interventions: Behavioral: isokinetic strength training of knee extensor and flexor muscles
- 5 assessments (Experimental): The randomisation provides for 5 assessments of baseline
  Interventions: Behavioral: isokinetic strength training of knee extensor and flexor muscles

INTERVENTIONS:
Behavioral: isokinetic strength training of knee extensor and flexor muscles — Patients underwent an isokinetic strength training program with 3 sessions per week during five weeks.
  Program consists of excentric contraction of knee flexor and extensor muscles (4 x 7 Contractions at 30°/s) and concentric contractions at maximal speed where patients can perform 40% of his maximal isometric torque for knee flexor and extensor muscles (2x10 for knee flexors and 2x10 for knee extensors)

SUMMARY:
The purpose of this study is to assess the impact of an isokinetic strength training of knee flexor and extensor muscles on walking performance in hemiparetic patients with knee extension thrust.

DETAILED DESCRIPTION:
The study will be interventional single case experimental design (SCED) with multiple baseline design. SCED are experimental designs aiming at testing the effect of an intervention using a small number of patients using repeated measurements, sequential and randomized introduction of an intervention and method-specific data analysis, including visual analysis and specific statistics.

During baseline, patients will have a rehabilitation program in day hospital (4 days per week) with physiotherapy and physical activity and if necessary occupational and speech therapy. Isokinetic strength training will be added to this conventionnal rehabilitation program and will begin after 3, 4 or 5 weeks of baseline according to randomization

12 patients will be included in this study (6 patients in subacute stage and 6 in chronic stage ).

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic patient (hemorragic or ischemic stroke)
* Subacute stage (< 6 Months) ou chronic stage of stroke (> 6 months) (6 patients in each group)
* Age between 18 and 75 years
* Able to walk 10 meters independently without any assistive devices
* Knee extension thrust during stance phase of gait cycle (rapid posterior movement of the knee toward extension)
* Scheduled rehabilitation program with isokinetic strength training
* affiliation to a social security
* Patients who received and signed informed consent

Exclusion Criteria:

* Major comprehension deficit that not allow to give informed consent and participate to isokinetic strength training (assessed with comprehension subscore of Langague screening Test)
* non stable (unstable cardiovascular condition)
* musculoskeletal disorders with knee pain that not allowed isokinetic strength training
* Botulinum toxin injection less than 3 months or repeated injection in lower limb,
* Proprioception trouble assessed with proprioception section of the Fugl-Meyer Assessment [FMA-P] 0/2
* spasticity of triceps surae ≥2 (Modified Ashworth scale)
* ankle dorsiflexion angle less than 90°
* pregnant women or breastfeeding
* persons with safety measure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
spontaneous walking speed | 25 weeks
  Spontaneous walking speed of hemiparetic patients recorded with 3D gait analysis

SECONDARY OUTCOMES:
Extensor thrust analysis | 25 weeks
  Extensor thrust at spontaneous and maximal walking speed and during dual task recorded with 3D gait analysis
Walking speed | 25 weeks
  assessment of walking speed in two conditions (maximal speed and dual task)
Stairs test | 25 weeks
  time to ascend and descend stairs (maximal speed)
Inclined plan | 25 weeks
  time to walk in an inclined plan (maximal speed)
6-minute walk test | 25 weeks
  Assessment of maximum gait perimeter during a 6MWT (6-minute walk test :6MWT)
Sit to stand test | 25 weeks
  1 minute sit to stand test (number of repetitions)
Extensor thrust during locomotor tasks | 25 weeks
  Extensor thrust analysis with inertial measurement unit (stairs, inclined walk, 6MWT and sit to stand )
Fatigue | 25 weeks
  Fatigue severity scale : FSS (minimum 9 -maximum 63 ; a higher score means higher level of fatigue)
Likert Scale | 25 weeks
  self perception of walking stability, fear of fall, trouble with extensor thrust with a likert scale
Strength | 25 weeks
  strength of knee flexor and extensor muscles assessed with isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Sophie HAMEAU, PhD, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France